CLINICAL TRIAL: NCT01480531
Title: Pre and or Post Operative Blood Pressure Control With Clevidipine (Cleviprexm Medicines Company) in Aortic Aneurysm / Dissection.
Acronym: Clevidipine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We elected to stop this study due to our inability to recruit suitable subjects.
Sponsor: Duke University (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030060
Record Dates: First submitted 2011-10-14; First posted 2011-11-29 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Aorta Aneurysm; Dissection of Aorta
Keywords: aorta; aneurysm; dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aneurysm | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevidipine — Clevidipine administration begins in the ER or ICU
  * Clevidipine is again administered post op when blood pressure control is required.
  * Clevidipine will be administered by an infusion pump via either a central line or a peripheral IV as follows:
  * Clevidipine will be initiated at an infusion rate of 0.4 μg•kg-1•min-1 and will be titrated as tolerated in doubling increments every 90 s up to 3.2 μg•kg-1•min-1.
  * Infusion rates above 3.2 μg•kg-1•min-1 will be guided by the patient's response and permitted in serial increments of 1.5 μg•kg-1•min-1.
  * Infusion rates between 4.4 and 8.0 μg•kg-1•min-1 will be administered for no longer than 2 h.
  As blood pressure approaches goal, increase dose by less than double and lengthen time between does adjustments to every 5-10 minutes (a 1-2 mg/hr increase will generally result in a 2-4 mm Hg reduction in SBP)
  Other Names: Cleviprex

SUMMARY:
2. Purpose of the Study -

1. To determine the feasibility of Clevidipine use for rapidly achieving and maintaining individually specified patient BP target ranges in the pre and postoperative periods of aortic aneurysm and dissection management.
2. To determine the safety of Clevidipine use in the pre and postoperative periods of aneurysm and dissection management
3. Background & Significance - Surgical treatments for persons with aortic root/arch dissection or aneurysm have significantly improved survival. However, critical in management of these patients is precise control of blood pressure (BP). With increasing BP, both acute and chronic, the risk of fatal and nonfatal vascular complications is imminent. Similarly, with excessive lowering of arterial pressures, cerebral, spinal cord, cardiac, and renal ischemic hypoperfusion is also noteworthy. Typically, the target systolic blood pressure range for these patients is 100-120 mmHg.

   Several different classes of vasoactive agents are in current use to acutely manage BP but none possess the optimal profile of an ideal vasodilator. Notable limitations include inadequate potency, slow onset and offset of action, multiple receptor function, safety concerns and, importantly, restricted/ineffective titration, which results in clinically significant hemodynamic and cardiovascular perturbations.

   Recently, the ultra short-acting intravenous dihydropyridine calcium-channel blocker clevidipine (Cleviprex, The Medicines Company) was approved for management of BP in critical care settings.

   Clevidipine's pharmacology lends itself to acute management of BP in a broad critical care setting in both surgical and nonsurgical patients. In the current study, the investigators propose to further characterize the hemodynamic effect of CLV in the pre and post-operative management of BP in patients with aortic aneurysm/dissection.
4. Design & Procedures Eligible patients will be approached to participate in the study by the Intensive Care Unit (ICU) attending and/or by a cardiothoracic surgical/anesthesiology fellow or a cardiac research nurse. All aspects of clinical management and monitoring will be according to standard practice that includes:

   * ECG
   * Oxymetry
   * Temperature
   * Invasive arterial blood pressure
   * Recording of routine laboratory results
   * Imaging studies including CT/MRI (A)/ Echocardiography
   * Pulmonary artery catheter (postoperative patients)
   * Mechanical ventilation (postoperative patients)
   * According to established protocol for acute intravenous management of arterial blood pressure in these patients, an upper and lower threshold of systolic blood pressure will be prescribed by the attending physician (the range being (100 mmHg -120 mm Hg SBP).

Hemodynamic data will be collected continuously via a bedside laptop as well as pertinent clinical data and information about efficacy and safety will be recorded.

• Subjective evaluation of efficacy of CLV (questionnaire format to be completed by the critical care team)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age 18-80 years)
2. Able to provide written consent
3. Type I and Type II (Type A) aortic dissection or unstable chronic aortic aneurysm
4. Patients expected to be admitted to ICU following aortic surgery for either dissection or aneurysm requiring acute management of elevated systolic blood pressure (consent obtained preoperatively)

Exclusion Criteria:

1. Unstable emergent dissections
2. Evidence of end-organ dysfunction (ischemia of spinal cord, bowel, myocardium or renal)
3. Active bleeding
4. Allergies to soybeans, soy products, eggs, or egg products; defective lipid metabolism such as pathologic hyperlipemia, lipoid nephrosis, or acute pancreatitis
5. Women who are pregnant
6. Female subjects of child bearing potential must have a blood serum pregnancy test performed prior to participating in this study and the results must be negative.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The use of Clevidipine to maintain clinically acceptable blood pressure. | Begining 24 hours prior to surgery thru 24 hours after surgery
  To determine the feasibility of Clevidipine use for rapidly achieving and maintaining individually specified patient BP target ranges (75 to 135 mm Hg) in the pre and postoperative periods of aortic aneurysm and dissection management.

SECONDARY OUTCOMES:
The incidence of hypotension | Begining 24 hours prior to surgery thru 24 hours after surgery
  To determine the safety of Clevidipine use in the pre and postoperative periods of aneurysm and dissection management to prevent hypotension as defined by a systolic blood pressure of less than 75 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Fontes, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Ericsson H, Fakt C, Hoglund L, Jolin-Mellgard A, Nordlander M, Sunzel M, Regardh CG. Pharmacokinetics and pharmacodynamics of clevidipine in healthy volunteers after intravenous infusion. Eur J Clin Pharmacol. 1999 Mar;55(1):61-7. doi: 10.1007/s002280050594. PMID 10206087
- [Background] Ericsson H, Fakt C, Jolin-Mellgard A, Nordlander M, Sohtell L, Sunzel M, Regardh CG. Clinical and pharmacokinetic results with a new ultrashort-acting calcium antagonist, clevidipine, following gradually increasing intravenous doses to healthy volunteers. Br J Clin Pharmacol. 1999 May;47(5):531-8. doi: 10.1046/j.1365-2125.1999.00933.x. PMID 10336577
- [Background] Bailey JM, Lu W, Levy JH, Ramsay JG, Shore-Lesserson L, Prielipp RC, Brister NW, Roach GW, Jolin-Mellgard A, Nordlander M. Clevidipine in adult cardiac surgical patients: a dose-finding study. Anesthesiology. 2002 May;96(5):1086-94. doi: 10.1097/00000542-200205000-00010. PMID 11981147
- [Background] Pollack CV, Varon J, Garrison NA, Ebrahimi R, Dunbar L, Peacock WF 4th. Clevidipine, an intravenous dihydropyridine calcium channel blocker, is safe and effective for the treatment of patients with acute severe hypertension. Ann Emerg Med. 2009 Mar;53(3):329-38. doi: 10.1016/j.annemergmed.2008.04.025. Epub 2008 Jun 5. PMID 18534716
- [Background] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012
- [Background] Aronson S, Boisvert D, Lapp W. Isolated systolic hypertension is associated with adverse outcomes from coronary artery bypass grafting surgery. Anesth Analg. 2002 May;94(5):1079-84, table of contents. doi: 10.1097/00000539-200205000-00005. PMID 11973166
- [Background] Reich DL, Bennett-Guerrero E, Bodian CA, Hossain S, Winfree W, Krol M. Intraoperative tachycardia and hypertension are independently associated with adverse outcome in noncardiac surgery of long duration. Anesth Analg. 2002 Aug;95(2):273-7, table of contents. doi: 10.1097/00000539-200208000-00003. PMID 12145033
- [Background] Weiss SJ, Longnecker DE. Perioperative hypertension: an overview. Coron Artery Dis. 1993 May;4(5):401-6. doi: 10.1097/00019501-199305000-00002. No abstract available. PMID 8261215
- [Background] Charlson ME, MacKenzie CR, Gold JP, Ales KL, Topkins M, Shires GT. Intraoperative blood pressure. What patterns identify patients at risk for postoperative complications? Ann Surg. 1990 Nov;212(5):567-80. doi: 10.1097/00000658-199011000-00003. PMID 2241312
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Vuylsteke A, Feneck RO, Jolin-Mellgard A, Latimer RD, Levy JH, Lynch C 3rd, Nordlander ML, Nystrom P, Ricksten SE. Perioperative blood pressure control: a prospective survey of patient management in cardiac surgery. J Cardiothorac Vasc Anesth. 2000 Jun;14(3):269-73. PMID 10890479
- [Background] Viljoen JF, Estafanous FG, Tarazi RC. Acute hypertension immediately after coronary artery surgery. J Thorac Cardiovasc Surg. 1976 Apr;71(4):548-50. PMID 817089
- [Background] Cheung AT, Cruz-Shiavone GE, Meng QC, Pochettino A, Augoustides JA, Bavaria JE, Ochroch EA. Cardiopulmonary bypass, hemolysis, and nitroprusside-induced cyanide production. Anesth Analg. 2007 Jul;105(1):29-33. doi: 10.1213/01.ane.0000264078.34514.32. PMID 17578949
- [Background] Aronson S, Fontes ML, Miao Y, Mangano DT; Investigators of the Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Risk index for perioperative renal dysfunction/failure: critical dependence on pulse pressure hypertension. Circulation. 2007 Feb 13;115(6):733-42. doi: 10.1161/CIRCULATIONAHA.106.623538. Epub 2007 Feb 5. PMID 17283267